CLINICAL TRIAL: NCT00231322
Title: The Influence of Transmission Season on Outcome of Schistosoma Haematobium Infection Treatment Among School Children in Urban and Peri-Urban Areas of Maputo and Matola, Mozambique
Brief Title: Influence of Transmission Season on Outcome of Treatment of Schistosoma Haematobium Infection in Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Durban University of Technology (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30/CNSB/03/624-03-0021
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Hematuria; Hydronephrosis
Keywords: Schistosoma haematobium; haematuria; ultrasonography; Uganda; Vesical polyps
MeSH Terms: conditions — Hematuria; Hydronephrosis; Schistosomiasis haematobia | interventions — Praziquantel

INTERVENTIONS:
Drug: praziquantel

SUMMARY:
To assess the influence of seasonal variations in Schistosoma haematobium transmission on treatment outcome (morbidity and re-infection)

DETAILED DESCRIPTION:
General objective To provide knowledge about the influence of transmission season (high and low) on the outcome of treatment assessed by cure rate, re-infection rate, regression and reappearance of urinary tract morbidity rate after treatment in order to optimise praziquantel treatment strategies for morbidity control in urinary schistosomiasis.

Specific objectives To determine the prevalence and intensity of Schistosoma haematobium infection before chemotherapy and compare cure rates and levels of re-infection after chemotherapy administered during high and low transmission seasons.

To assess urinary tract morbidity due to Schistosoma haematobium by ultrasonography and compare the regression and reappearance of urinary tract pathology chemotherapy administered during high and low transmission seasons.

To correlate morbidity determined by ultrasound with infection and morbidity parameters such as intensity of infection, micro- and macrohematuria, circulating cathodic antigen (CCA) in urine, proteinuria and leucocyturia and determine sensitivity, specificity and positive predictive values in relation to urinary tract morbidity.

Study design The main research question concerning the influence of transmission season on treatment outcome will be addressed in a consecutive cohort study with two separate but comparable cohorts. The first cohort will be examined and treated with praziquantel during the season with high transmission, February/Mach (group A) and the second cohort will be examined and treated during the low transmission season, in July approximately 5 months later (group B). Each cohort will be examined before treatment and 2, 6 and 18 months after treatment.

The study will be carried out in 4 primary schools; two from Machava J area and two from Costa do Sol area. The schools will be selected based on the following criteria: similar prevalence (> 50%) and intensity of S. haematobium infection; absence or very low levels of S. mansoni infection; a minimum of 2 classes (>35 pupils per class) at each level (3rd and 4th level) and similar distribution of boys and girls.Examinations will include urine for parasitology and haematuria and ultrasonography of upper and lower urinary tract

ELIGIBILITY:
Inclusion Criteria:

* children aged 8-12 years

Exclusion Criteria:

* All children presenting with macro-haematuria or severe pathology detected by ultrasonography (large masses, pseudo-polyps or hydronephrosis/hydroureter) at the 6 months follow-up examination will be treated with praziquantel and excluded in the data analysis.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520
Dates: Start 2004-03; Study Completion 2006-03

PRIMARY OUTCOMES:
cure rate
egg reduction rate
re-infection prevalence and intensity of infection *resolution of urinary tract pathology
re-appearance of pathology after re-infection.

SECONDARY OUTCOMES:
reduction in worm burden (CAA);

CONTACTS AND LOCATIONS:
Overall Officials: Gerito Augusto, Msc, Principal Investigator — Instituto Nacional de Saúde, Mozambique
Locations (1):
- Matola, Maputo, Maputo Province, Mozambique

REFERENCES:
- See also: Related Info — http://www.dblnet.dk